CLINICAL TRIAL: NCT02217163
Title: Study of Carfilzomib in Transplant Eligible Newly Diagnosed High-risk Multiple Myeloma
Brief Title: Carfilzomib, Cyclophosphamide, Dexamethasone in Transplant Eligible Newly Diagnosed High-risk Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGHMM1
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): The combination therapy of Carfilzomib, cyclophosphamide and dexamethasone (KCyd) will be used to treat eligible patients for up to 6 cycles.This will be followed by an autologous bone marrow transplantation and 2 further consolidation cycles of KCyd. Depending on their disease response, patients will be managed expectantly or be started on maintenance.
  Interventions: Drug: Carfilzomib, , Cyclophosphamide, Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib, , Cyclophosphamide, Dexamethasone — Carfilzomib is administered intraveneously over 30 minutes. For cycle 1 only, Carfilzomib is administered at 20mg/m2 on Day 1 and 2, dose will be escalated to 36mg/m2 on Day 8,9,15 and 16 of the 28-days cycle. Patients who tolerate the 36mg/m2 dose are kept at this dose for the subsequent cycles on Day 1,2,8,9,15,16 on a 28 days cycle. Cyclophosphamide is given at a fixed dose of 500mg once per week orally, along with dexamethasone which is given on the days of Carfilzomib administration, 30 minutes to 4 hours prior to Carfilzomib infusion.
  Other Names: Kyprolis

SUMMARY:
Patients with high risk multiple myeloma have shorter remission periods and reduced overall survival. Prognostic significance of minimal residual disease negative remission is being highlighted in many of the newer studies.

The current phase 2 study investigates the combination of carfilzomib together with cyclophosphamide and dexamethasone in patients with high risk multiple myeloma in younger transplant-eligible patients.

DETAILED DESCRIPTION:
Carfilzomib is administered over 30 minutes as an infusion. For cycle 1 only, Carfilzomib is administered at 20mg/m2 IV on days 1 and 2, followed by escalation to 36 mg/m2 on days 8,9,15 and 16 on a 28 day cycle. Patients who tolerate 36 mg/m2 dose are kept at this dose for the subsequent cycles on Days 1, 2, 8, 9, 15, 16 on a 28 day cycle. Dose and schedule modifications for intolerable side effects are detailed in the protocol. Additionally Cyclophosphamide is given a fixed dose of 500mg once per week orally, along with dexamethasone, given on the days of Carfilzomib administration, 30 minutes to 4 hours prior to Carfilzomib. Patients will undergo blood tests weekly and serum protein electrophoresis every 4 weeks during treatment. Within completion of 5 cycles of treatment, patients would undergo stem cell collection using chemotherapy and GCSF mobilization. After completion of 6 cycles of treatment, autologous bone marrow transplantation will be performed. Three months following bone marrow transplantation, subjects will undergo further 2 consolidation cycles. After consolidation, subjects will undergo disease assessment by blood and subjects who are in CR will undergo bone marrow investigations and MRD analysis MPFC. Patients who achieve MRD negativity by MPFC will be managed expectantly by watch and wait. Patients who are MRD positive at this stage will receive maintenance for 2 years or till disease progression. Follow up would extend till a minimum of 2 years from completion of the study. At the end of 2 years post maintenance or expectant monitoring, subjects who are in CR will undergo disease assessment by blood and bone marrow investigations and MRD analysis MPFC.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed Multiple Myeloma AND Transplant eligible AND
2. High Risk as defined by:

   * International Staging System 3 OR
   * FISH abnormality of t(4,14), t(14;16), 17p deletion or 1q amp
3. Patients must have evaluable myeloma, with at least one of the following (Assessed within 28 days of commencing the study)

   * Serum M protein >/= 0.5g/dL or
   * Urine M protein >200mg/24hr
   * Serum free light chains >100mg/mL (involved light chain) and abnormal k/l ratio
   * For IgA patients who have no other means of measurement of disease, sIgA level >0.75g/dL

Exclusion Criteria:

1. Relapsed Myeloma
2. Non transplant eligible patient.
3. IgM subtype Myeloma
4. POEMS syndrome
5. Amyloidosis
6. Waldenstroms Macroglobulinemia
7. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days of randomization (Limited site radiation allowed).

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years
  To study the progression free survival (PFS) in patients with newly diagnosed high risk multiple myeloma treated with Carfilzomib, Cyclophosphamide and Dexamethasone, followed by autologous bone marrow transplantation.

SECONDARY OUTCOMES:
Minimal residual disease negativity | 2 years
  Minimal residual disease burden at different time points, as assessed by multi parameter flow cytometry (MPFC).
Overall Survival (OS) | 2 years
  OS is defined as the time from entering study to death of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Chandramouli Nagarajan, MBBS, Principal Investigator — Singapore General Hospital
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore